CLINICAL TRIAL: NCT04829656
Title: Identifying Factors Predicting ACcurately End-of-Life in Dementia With Lewy Bodies and Promoting Quality End-of-Life Experiences: the PACE-DLB Study
Brief Title: The PACE-DLB Study
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB202001438; 1R01AG068128-01 (NIH)
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Dementia With Lewy Bodies
Keywords: dementia; Lewy bodies; Lewy body; aging; neurology
MeSH Terms: conditions — Lewy Body Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Cohort: Enrolled via the 5 participating clinics at LBDA Research Centers of Excellence.
- Virtual Cohort: Enrolled via the LBDA.

SUMMARY:
The PACE-DLB Study is for people with at least moderate dementia with Lewy bodies (DLB) and their primary caregiver. The study's goals are to learn more about the experiences of people with DLB and their caregivers as DLB progresses, and what happens as the end of life of the person with DLB approaches. Participants are enrolled through one of five Lewy Body Dementia Association (LBDA) Research Center of Excellence clinics, or directly via the LBDA.

People with DLB will enroll into the study along with their primary informal caregiver, such as the family member or friend who is involved in most of their care and attends the majority of their medical appointments. A legally authorized representative (LAR) for the person with DLB will consent to participate in the study on the person's behalf. If the person with DLB resists taking part in the study, the pair will not be enrolled.

The study consists of questionnaires about the progression of the person's dementia and the experiences of the caregiver. The person with DLB will complete one questionnaire themselves if they are able to. If the pair is enrolled at a LBDA Research Center of Excellence clinical site, and completes study visits in-person, a brief physical exam of the person with DLB will be completed by a clinician.

Study participation will last for three years, or until the person with DLB dies. Study visits take place every six months, either virtually or in person at a clinical study site. If the person with DLB dies during the study, the caregiver will complete one final virtual study visit three months afterward.

Specific Aims of the PACE-DLB Study:

1. To determine predictors of the end of life (death within 6 months) in the DLB population.

   Hypotheses: Predictors of death within 6 months for individuals with DLB will include symptoms (e.g. worsening hallucinations, fluctuations) not captured in existing dementia end-of-life prediction tools.
2. To identify whether change in caregiver measures can predict the end of life in the DLB.

   Hypotheses: The investigators hypothesize that there will be worsening caregiver burden, depression, grief, and quality of life preceding the last 6 months of life, controlling for variables such as resilience, support, and living situation.
3. To identify the impact of demographics, health care factors, and specific DLB symptoms on patient quality of life and caregiver experiences at the end of life of the person living with DLB.

Hypotheses: Location (rural, urban, suburban), provider experience (e.g. specialist vs not), patient residence (e.g. home, skilled nursing), degree of behavioral symptoms, caregiver type (spouse vs child vs other), and caregiver characteristics (self-efficacy, perceived social support, resilience, and coping) will affect patient and informal caregiver experiences at the patient's end of life, including patient and caregiver quality of life and caregiver well-being, depression, burden, grief, and satisfaction with end-of-life care.

DETAILED DESCRIPTION:
Dementia with Lewy bodies (DLB) is part of Lewy body dementia, the 2nd-most-common degenerative dementia in the U.S. It is also one of the Alzheimer's disease-related dementias (ADRDs). Evidence-based models of end-of-life care for ADRDs are insufficient; families face difficult medical decisions with little information for guidance. This is particularly relevant for DLB, where >70% of individuals die of the dementia itself or failure to thrive. Caregivers describe lack of knowledge of what to expect at the end of life as an important driver of negative end-of-life experiences. The proposed study addresses this unmet need. It also addresses the National Institute on Aging's priority to improve quality of care and quality of life for persons with ADRDs at the end of life and their caregivers.

Based on published clinical series, over half of enrolled individuals with DLB are expected to die over the course of the study. To achieve diverse recruitment, the study includes an in-person cohort where dyads are recruited from Lewy Body Dementia Association Research Centers of Excellence and a novel virtual cohort where dyads are recruited through the Lewy Body Dementia Association and study visits are conducted by telephone. Having a virtual cohort will capture the experiences of individuals with DLB and caregivers not receiving care at specialty centers.

Because the majority of study measures are caregiver-reported, the in-person and virtual groups have identical study measures, except for the Unified Parkinson Disease Rating Scale, completed only in person. Collected measures will include demographics, DLB characteristics (e.g. cognitive, motor, behavioral, sleep, and autonomic symptoms), health care providers and settings, caregiver considerations (e.g. resilience, support, grief, burden), quality of life (for the patient and caregiver), and satisfaction with end of life experiences.

The caregiver will complete a final study visit 3 months after the death of the person with DLB to assess grief, recovery, and quality of the end of life experience. By following dyads through the end of life and death of the person with DLB and the initial bereavement period for the caregiver, the study will identify DLB-specific predictors of the last 6 months of life, changes in caregiver measures that identify the last 6 months of life, and factors which influence quality end of life experiences. These results will inform the content and timing of end-of-life counseling in DLB, help establish quality metrics for end of life care, and identify areas where interventions could potentially improve end of life experiences for individuals with DLB and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patient and caregiver willing to participate as a dyad (patients will need a legally authorized representative to consent on their behalf given the requirement for at least moderate dementia, but patients who resists participating in the study will not be enrolled)
* U.S. residents (i.e., individuals accessing the LBDA from outside the U.S. will be excluded)
* Patient with a clinical diagnosis of DLB
* Patient with moderate severity dementia as assessed by the Quick Dementia Rating System (QDRS, with a score of >12 OR ≥2 in at least 3 domains suggestive of moderate dementia)
* Caregiver telephone interview for cognitive status (TICS) score of >31 to ensure that the caregiver is able to reliably complete study visits
* Patient participant expected to live at least 6 months (so that at least a baseline visit and 1 follow up visits is expected to be completed)

Exclusion Criteria:

* Patient participant diagnosed with dementia of less than moderate severity
* Patient with dementia resists participation
* Non-U.S. residents
* Patient participant with dementia not expected to live at least 6 months
* Virtual cohort ONLY: Patient participant receives medical care from a LBDA Research Centers of Excellence clinic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at five LBDA Research Centers of Excellence clinics may enroll into the study if they meet inclusion criteria. Clinics participating in the study are located at the University of Florida, Gainesville, FL; University of Miami, Miami, FL; University of Virginia, Charlottesville, VA; University of Michigan, Ann Arbor, MI; and the Mayo Clinic, Rochester, MN.
  People who have indicated interest in research opportunities through the LBDA mailing listserv will be emailed study information, including how to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Predictors of the end of life (death within 6 months) in the DLB population | Every 6 months for up to 3 years
  The investigators define a variable that predicts the end of life as a variable changing substantially (e.g., quick drop of quality of life) once the patient enters last six months of life. The investigators will model and estimate the longitudinal trajectories of all potential candidate variables to identify those with significantly different trajectory patterns in the last six months of life.
Identify whether change in caregiver measures can predict the end of life in the DLB | Every 6 months for up to 3 years
  The investigators will collect caregiver measures such as quality of life, burden, depression, dementia-related grief, support, resilience, and coping for all dyads (virtual and clinical cohorts). The investigators will assess the correlation between (1) caregiver burden, depression, grief, and quality of life scores and (2) change in caregiver burden, depression, grief, and quality of life scores with the last 6 months of life of the person with DLB.
Identify the impact of demographics with specific DLB symptoms on patient quality of life and caregiver experiences at the end of life of the person living with DLB | Every 6 months for up to 3 years
  Using both the virtual and clinical cohorts, the investigators will identify which patient demographics (e.g. age, gender, sex, race/ethnicity, disease duration, level of education), caregiver demographics (e.g. age, gender, sex, race/ethnicity, relationship to patient, level of education), disease characteristics (e.g. overall symptom burden, cognition, motor function, neuropsychiatric symptoms, functional status, fluctuations, sleep-related symptoms, autonomic symptoms, medications), elements of care (rural/urban, type of healthcare provider, patient residence), and caregiver measures (self-efficacy, social support, coping skills) drive patient (QoL) and caregiver (QoL, depression, burden, grief, resilience) outcomes. These will be assessed across the disease course and specifically at the end of life (at the last clinical visit prior to death).

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Armstrong, MD, MSc, FAAN, Principal Investigator — University of Florida
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Armstrong MJ, Wollney E, Li Z, Dai Y, LaBarre B, Wang T, Sovich K, Jury HF, Galvin JE, Henriquez AM, Maixner SM, Paulson HL, Fields JA, Lunde A, Boeve BF, Manning C, Taylor AS, Baker ZG. Caregiver experiences after the death of a person with dementia with Lewy bodies: A mixed-methods analysis. J Alzheimers Dis. 2025 Oct;107(3):1097-1113. doi: 10.1177/13872877251365218. Epub 2025 Aug 14. PMID 40808538
- [Derived] Wollney E, Sovich K, LaBarre B, Maixner SM, Paulson HL, Manning C, Fields JA, Lunde A, Boeve BF, Galvin JE, Taylor AS, Li Z, Fechtel HJ, Armstrong MJ. End-of-life experiences in individuals with dementia with Lewy bodies and their caregivers: A mixed-methods analysis. PLoS One. 2024 Aug 29;19(8):e0309530. doi: 10.1371/journal.pone.0309530. eCollection 2024. PMID 39208192
- [Derived] Armstrong MJ, Dai Y, Sovich K, LaBarre B, Paulson HL, Maixner SM, Fields JA, Lunde AM, Forsberg LK, Boeve BF, Manning CA, Galvin JE, Taylor AS, Li Z. Caregiver Experiences and Burden in Moderate-Advanced Dementia With Lewy Bodies. Neurol Clin Pract. 2024 Jun;14(3):e200292. doi: 10.1212/CPJ.0000000000200292. Epub 2024 Apr 10. PMID 38617555
- [Derived] Armstrong MJ, LaBarre B, Sovich K, Maixner SM, Paulson HL, Manning C, Fields JA, Lunde A, Forsberg L, Boeve BF, Galvin JE, Taylor AS, Li Z. Patient- and proxy-reported quality of life in advanced dementia with Lewy bodies. Alzheimers Dement. 2024 Apr;20(4):2719-2730. doi: 10.1002/alz.13745. Epub 2024 Feb 23. PMID 38400528
- [Derived] Armstrong MJ, Paulson HL, Maixner SM, Fields JA, Lunde AM, Boeve BF, Manning C, Galvin JE, Taylor AS, Li Z. Protocol for an observational cohort study identifying factors predicting accurately end of life in dementia with Lewy bodies and promoting quality end-of-life experiences: the PACE-DLB study. BMJ Open. 2021 May 26;11(5):e047554. doi: 10.1136/bmjopen-2020-047554. PMID 34039578